CLINICAL TRIAL: NCT04270695
Title: Effects of Blood Flow Restriction Training Combined With Abdominal draw-in Maneuver on Transverse Abdominis Strengthening
Brief Title: Blood Flow Restriction Training Combined With Abdominal draw-in Maneuver on Transverse Abdominis Strengthening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Yueh-Ling Hsieh, professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CRREC-109-007
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-10

CONDITIONS: Blood Flow Restriction; draw-in Maneuver; Transverse Abdominis
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blood flow restriction (Experimental): An inflatable cuff (14 cm in width * 84 cm in length) is warped around abdominal muscles below ribs which may cause to at least 60% restriction of blood flow detected by Power Doppler ultrasonography. All participants are instructed to perform abdominal draw-in maneuver both condition of BFR and BFR-free twice a week, for six weeks.
  Interventions: Behavioral: blood flow restriction
- sham blood flow restriction (Sham Comparator): an inflatable cuff (14 cm in width * 84 cm in length) is warped around abdominal muscles below ribs without inflation. All participants are instructed to perform abdominal draw-in maneuver.
  Interventions: Behavioral: sham blood flow restriction

INTERVENTIONS:
Behavioral: blood flow restriction — an inflatable cuff (14 cm in width * 84 cm in length) is warped around abdominal muscles below ribs which may cause to at least 60% restriction of blood flow detected by Power Doppler ultrasonography. All participants are instructed to perform abdominal draw-in maneuver.
  Arms: blood flow restriction
Behavioral: sham blood flow restriction — an inflatable cuff (14 cm in width * 84 cm in length) is warped around abdominal muscles below ribs without inflation. All participants are instructed to perform abdominal draw-in maneuver.
  Arms: sham blood flow restriction

SUMMARY:
This study expects to provide a new alternative way to improve the muscle activation, strength and activation of transverse abdominis in abdominal draw-in maneuver combined with blood flow restriction.

DETAILED DESCRIPTION:
The transverse abdominis (TrA) is the deepest muscle layer of lateral and anterior abdominal wall and also known as a significant component of core stability. Abdominal draw-in maneuver (ADIM) is the main for the strengthening of the deep muscle, however, sufficient activation of TrA by ADIM is limited. Blood flow restriction (BFR) training is a technique combined with low intensity exercise that produces similar results to high intensity training. However, there is few evidences for BFR training on core muscles.

Healthy adults (age ranged 18-34 years and BMI between 18.5~24.99) were randomly recruited in the study. For the intervention group, an inflatable cuff (14 cm in width * 84 cm in length) is warped around abdominal muscles below ribs which may cause to at least 60% restriction of blood flow detected by Power Doppler ultrasonography. All participants are instructed to perform ADIM both condition of BFR and BFR-free twice a week, for six weeks. Outcome measurements include Double leg lowering test (DLLT) for muscle strength, brightness mode ultrasound (USD) for muscle hypertrophy and electromyography (EMG) muscle activation. The same physical therapist will do the measurement at first week, third week and the sixth week.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* 20~35 years old
* BMI 18.5~24.99

Exclusion Criteria:

* Hypertension
* Have cardio-vascular disease
* Used to have abdominal operation or wound
* Have spinal surgeries or deformities
* Known neuromuscular or joint disease
* Pregnant

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-04-03 (Actual); Study Completion 2021-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Ling Hsieh, Study Director — professor
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: participants were recruited from college aged between 20~35
Pre-assignment Details: of 37 participants, 36 met the inclusion criteria while 1 participant was excluded because of overweighted.
Groups:
- Blood Flow Restriction: An inflatable cuff (14 cm in width * 84 cm in length) is warped around abdominal muscles below ribs and inflated to 160mm-Hg which may cause to at least 60% restriction of blood flow detected by Power Doppler ultrasonography. All participants are instructed to perform abdominal draw-in maneuver in condition of BFR twice a week, for six weeks.
  blood flow restriction: an inflatable cuff (14 cm in width * 84 cm in length) is warped around abdominal muscles below ribs which may cause to at least 60% restriction of blood flow detected by Power Doppler ultrasonography. All participants are instructed to perform abdominal draw-in maneuver.
- Sham Blood Flow Restriction: An inflatable cuff (14 cm in width * 84 cm in length) is warped around abdominal muscles below ribs without inflation as a sham operation.All participants are instructed to perform abdominal draw-in maneuver in condition of BFR-free twice a week, for six weeks.
Period: Overall Study
Arm/Group | Blood Flow Restriction | Sham Blood Flow Restriction
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blood Flow Restriction | Sham Blood Flow Restriction | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.47 (1.33) | 21.53 (1.69) | 21.5 (1.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 7 | 9 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 17 | 17 | 34
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21.41 (0.93) | 21.53 (1.69) | 21.5 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Muscle Thickness Change of Transverse Abdominis
Description: muscle thickness change on week3, 4 and 5 compared with baseline
Time Frame: 3,4,5 weeks
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Blood Flow Restriction: wrap an inflatable cuff below the 12 ribs and inflated to 160 mmHg
- Sham Blood Flow Restriction: wrap an inflatable cuff below the 12 ribs but deflated
Arm/Group | Blood Flow Restriction | Sham Blood Flow Restriction
Number analyzed (Participants) | 17 | 17
mm
  baseline | 0.93 (0.97) | 0.77 (1.45)
  week 3 | 1.98 (1.4) | 0.99 (0.79)
  week 4 | 2.65 (1.08) | 0.78 (0.79)
  week 5 | 2.7 (1.62) | 0.83 (0.75)

2. Secondary Outcome: Internal Oblique Thickness Change
Description: Data represents the muscle thickness change on week 3, 4 and 5 compared with baseline. The thickness of the muscle was calculated by the differences between the muscle thickness during contraction and the muscle thickness during resting position. If the muscle thickness during contraction was smaller than the muscle thickness during the resting position, therefore, the values would be negative. The values in baseline presented as negative may be because the internal oblique muscle thickness during contraction was smaller before receiving any training. Previous studies stated that after receiving ADIM and BFR training, the internal oblique muscle thickness will be thicker. Therefore, it was reasonable that the results in baseline presented negative values while the values became positive after receiving training.
Time Frame: baseline,3,4,5 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Blood Flow Restriction | Sham Blood Flow Restriction
Number analyzed (Participants) | 17 | 17
mm
  baseline | -0.01 (1.06) | -0.2 (1.09)
  week 3 | 0.75 (1.72) | 0.02 (1.04)
  week 4 | 0.96 (2.66) | 0.14 (0.94)
  week 5 | 1.21 (1.53) | 0.4 (1.78)

3. Secondary Outcome: External Oblique Thickness Change
Description: Data represents the muscle thickness change on week 3, 4 and 5 compared with baseline. The thickness of the muscle was calculated by the differences between the muscle thickness during contraction and the muscle thickness during resting position. If the muscle thickness during contraction was smaller than the muscle thickness during the resting position, therefore, the values would be negative. The values in baseline presented as negative may be because the external oblique muscle thickness during contraction was smaller before receiving any training. After receiving ADIM and BFR training, the tranverse abdominis and internal oblique muscle thickness will be thicker while the external oblique will be thinner due to the compression from the TrA and IO muscles.
Time Frame: baseline,3,4,5weeks
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Blood Flow Restriction: An inflatable cuff (14 cm in width * 84 cm in length) is warped around abdominal muscles below ribs and inflated to 160mm-Hg which may cause to at least 60% restriction of blood flow detected by Power Doppler ultrasonography. All participants are instructed to perform abdominal draw-in maneuver in condition of BFR twice a week, for five weeks.
  blood flow restriction: an inflatable cuff (14 cm in width * 84 cm in length) is warped around abdominal muscles below ribs which may cause to at least 60% restriction of blood flow detected by Power Doppler ultrasonography. All participants are instructed to perform abdominal draw-in maneuver.
- Sham Blood Flow Restriction: An inflatable cuff (14 cm in width * 84 cm in length) is warped around abdominal muscles below ribs without inflation as a sham operation.All participants are instructed to perform abdominal draw-in maneuver in condition of BFR-free twice a week, for five weeks.
Arm/Group | Blood Flow Restriction | Sham Blood Flow Restriction
Number analyzed (Participants) | 17 | 17
mm
  baseline | -0.77 (1.08) | -0.47 (1.04)
  week 3 | -0.97 (1.11) | -0.41 (0.76)
  week 4 | -0.94 (1.09) | -0.16 (0.8)
  week 5 | -0.95 (1.02) | -0.68 (1.13)

ADVERSE EVENTS:
Description: All Mortality, Serious, and Other Adverse Events (ex, injury )were not monitored/assessed
Arm/Group | Blood Flow Restriction | Sham Blood Flow Restriction
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT04270695/Prot_SAP_000.pdf